CLINICAL TRIAL: NCT02102503
Title: Motivational Interviewing and Medication Review in the Secondary Prevention of Coronary Heart Disease
Brief Title: Motivational Interviewing and Medication Review in Coronary Heart Disease
Acronym: MIMeRiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göran Petersson (Other)
Collaborators: The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other)
Responsible Party: Sponsor-Investigator, Göran Petersson, Professor of Health Informatics with focus on Pharmaceutical Science, Linnaeus University
Organization: Linnaeus University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GLAS-1-2013
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Medication Review

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI and Medication review (Experimental): The intervention starts three months post-discharge after the standard treatment at the out-patients clinic. A medication review focused on cardiovascular drugs, and a counselling session with a clinical pharmacist using Motivational Interviewing (MI)-approach, and a follow-up phone call two weeks later. For patients with negative beliefs about medicines, three additional MI-sessions in clinic or by phone are planned together with the patient. Irrespective of beliefs the intervention ends with a second medication review and counselling session, which is coordinated with the 12-months post-discharge follow-up in primary care.
  Interventions: Behavioral: Standard Treatment; Behavioral: MI and Medication review
- Standard treatment (Active Comparator): Standard treatment at the cardiology out-patient clinic. Follow-up by nurse after two weeks and by physician after two months.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Standard Treatment
Behavioral: MI and Medication review
  Arms: MI and Medication review

SUMMARY:
Low medication adherence in patients with coronary heart disease increases mortality.

This study investigates if an intervention of medication review and counselling can improve patients' medication adherence and treatment results.

DETAILED DESCRIPTION:
The study will investigate the effects of medication review and Motivational Interviewing (MI) on patients with Coronary Heart Disease (CHD). Clinical pharmacists competent in MI and cardiology will conduct medication interviews and medication reviews at the outpatient clinic. The intervention will continue during 9 months, with interviews and reviews as needed.

Follow-up of results will take place 16 months after inclusion (corresponding to 4 months after the end of intervention).

The MI-Component will be quality assured by MITI 4.2-coding (Motivational Interviewing Treatment Integrity). The study will investigate effects on clinical outcomes, medication adherence, patients´ beliefs about medicines and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for angiography
* Verified Coronary Artery Disease (ICD-10 I20-I21)
* Planned for follow up at the out-patient clinic (standard treatment)
* Swedish speaking

Exclusion Criteria:

* Cognitive impairment or any othe condition making interview or phone calls impossible.
* Non-participation in the standard follow-up
* Prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2013-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve the treatment goal for Low density lipoprotein cholesterol (LDL-C) | 16 months
  According to Swedish guidelines the goal is < 1,8mmol/L or at least 50% reduction from baseline.

SECONDARY OUTCOMES:
Percentage of patients adherent to cholesterol lowering treatment | 16 months
  Self-reported adherence according to Morisky-8-Item Adherence Scale
Percentage of patients adherent to cholesterol lowering treatment | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, 1 refill month 12-16 is set as the cut-off for adherence.
Percentage of patients adherent to cholesterol lowering treatment | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, Percent Day Covered (PDC) during follow-up period, 80% is set as the cut-off for adherence.
Percentage of patients adherent to preventive medication: Angiotensin Converter Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, 1 refill month 12-16 is set as the cut-off for adherence.
Percentage of patients adherent to preventive medication: Acetylsalicylic acid (ASA) | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, 1 refill month 12-16 is set as the cut-off for adherence.
Percentage of patients adherent to preventive medication: P2Y12-antagonist | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, 1 refill month 12-16 is set as the cut-off for adherence.
Percentage of patients adherent to preventive medication: Beta-blocker | 16 months
  Prescription refill according to the Swedish Prescribed Drug Register, 1 refill month 12-16 is set as the cut-off for adherence.
Percentage of patients with Systolic Blood Pressure <140 | 16 months
  As registered in the Electronic Health Record
Changes in Quality of Life | 16 months
  The Heart QoL instrument
Number of Cardiovascular Re-admissions and Emergency Department visits | 16 months
  According to the Health Care register of Kalmar County

OTHER OUTCOMES:
Process measure: Quality of prescribing, for a random sample of 20 % of patients | 6 months
  According to Medication Assessment Tool for secondary prevention of Coronary Heart disease
Process measure: What was delivered in the Medication review | 12 months, only intervention group
  Number and type of drug-related problems, as categorized by Cipolle and Strand. And documented effects of any actions taken on drug-related problems.
Process measure: Quality of MI, for a random sample of 20 % of consultations | 12 months
  According to MITI 4.2.1
Process measure: Beliefs about medicines - percent of patients per category | 16 months
  Beliefs about medicines questionnaire (BMQ-S10), categories: accepting, ambivalent, neutral, skeptical. Also temporal cahnges in both Groups and Changes in each item of the subscales.
Process measure: Intervention experienced by patients | 12 months
  Qualitative interview study of 8-15 patients with negative beliefs about medicines at baseline. Analyzed with content analysis.
Process measure: How did the intervention affect patients´overall experience of their follow-up care after CHD. | 16 months, for the last 100 patients to be included.
  Open question: What is you opinion of the follow-up care after your heart disease?" Analysed with qualitative content analysis separetly for Control and intervention group patients.
Health economic evaluation: Costs of intervention related to costs saved and Quality-adjusted Life years | 16 months
  Quality adjusted life years estimated by the re-admissions and quality of Life using Euroqol EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Göran Petersson, MD, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Kalmar County Hospital, Kalmar, Sweden

REFERENCES:
- [Derived] Ostbring MJ, Eriksson T, Petersson G, Hellstrom L. Effects of a pharmaceutical care intervention on clinical outcomes and patient adherence in coronary heart disease: the MIMeRiC randomized controlled trial. BMC Cardiovasc Disord. 2021 Aug 1;21(1):367. doi: 10.1186/s12872-021-02178-0. PMID 34334142
- [Derived] Ostbring MJ, Eriksson T, Petersson G, Hellstrom L. Motivational Interviewing and Medication Review in Coronary Heart Disease (MIMeRiC): Protocol for a Randomized Controlled Trial Investigating Effects on Clinical Outcomes, Adherence, and Quality of Life. JMIR Res Protoc. 2018 Feb 20;7(2):e57. doi: 10.2196/resprot.8659. PMID 29463490